CLINICAL TRIAL: NCT00074204
Title: A Phase III Study of Delayed vs. Immediate Second-Line Therapy With Docetaxel After Gemcitabine + Carboplatin in Advanced Non-Small Cell Lung Cancer
Brief Title: Gemcitabine and Carboplatin Followed By Docetaxel in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Nathan Levitan, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LILY1503; P30CA043703 (NIH); CASE-CWRU-LILY-1503 (Other: Case Comprehensive Cancer Center); LILLY-B9E-US-S245
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Docetaxel (Experimental): Arm I (immediate docetaxel): Patients receive immediate docetaxel IV over 1 hour on day 1.
  Interventions: Drug: carboplatin; Drug: docetaxel; Drug: gemcitabine hydrochloride
- Delayed Docetaxel (Active Comparator): Arm II (delayed docetaxel): Patients are observed until first evidence of disease progression and then receive docetaxel IV over 1 hour on day 1.
  Interventions: Drug: carboplatin; Drug: docetaxel; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: carboplatin — Carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
Drug: docetaxel — Arm I (immediate docetaxel): Patients receive immediate docetaxel IV over 1 hour on day 1.
  Arm II (delayed docetaxel): Patients are observed until first evidence of disease progression and then receive docetaxel IV over 1 hour on day 1.
  In both arms, treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Drug: gemcitabine hydrochloride — Gemcitabine IV over 30-60 minutes on days 1 and 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, carboplatin, and docetaxel, use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which treatment regimen is more effective for stage IIIB or stage IV non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of gemcitabine and carboplatin followed immediately by docetaxel with that of giving delayed docetaxel in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with stage IIIB or IV non-small cell lung cancer treated with gemcitabine and carboplatin followed by immediate vs delayed docetaxel.

Secondary

* Compare the response rate and time to progression in patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to ECOG performance status (0 or 1 vs 2).

All patients receive gemcitabine IV over 30-60 minutes on days 1 and 8 and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with stable or responding disease proceed to docetaxel therapy. Patients are randomized to 1 of 2 treatment arms.

* Arm I (immediate docetaxel): Patients receive immediate docetaxel IV over 1 hour on day 1.
* Arm II (delayed docetaxel): Patients are observed until first evidence of disease progression and then receive docetaxel IV over 1 hour on day 1.

In both arms, treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life (QOL) is assessed at baseline, at restaging (after completion of gemcitabine and carboplatin), before courses 2-6 of docetaxel*, and then at 1 and 3 months after study treatment.

NOTE: *For patients randomized to delayed docetaxel, QOL is assessed every 3 weeks until first disease progression and then before courses 2-6 of docetaxel

Patients are followed monthly for 3 months, every 2 months for 6 months, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 550 patients (275 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Stage IIIB with pleural effusion OR stage IV disease
  * Recurrent disease after primary treatment with radiotherapy or surgery allowed
* Measurable disease or nonmeasurable disease

  * Measurable disease, defined as at least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Nonmeasurable disease, defined as all other lesions, including small lesions (longest diameter less than 20 mm by conventional techniques OR less than 10 mm by spiral CT scan) or any of the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Cystic lesions
    * Abdominal masses not confirmed and followed by imaging techniques
* No symptomatic CNS metastases

  * Treated, stable CNS metastases allowed provided patient is not receiving radiotherapy or corticosteroids

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 3.0 times upper limit of normal (ULN) (less than 5.0 times ULN for patients with documented benign disease)
* Alkaline phosphatase less than 3.0 times ULN (for patients with documented benign disease)

Renal

* Creatinine no greater than 1.5 mg/dL

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study participation
* No active and ongoing infection
* No concurrent serious systemic disorder that would preclude study participation
* No other primary malignancy within the past 5 years except carcinoma in situ of the cervix, adequately treated basal cell skin cancer, or T1 vocal cord cancer in remission

  * Other prior cancers unlikely to affect survival for the next 3 years (e.g., low-grade early stage prostate cancer) are allowed

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No prior chemotherapy for NSCLC, including neoadjuvant and adjuvant therapy
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent antitumor hormonal therapy (excluding contraceptives and replacement steroids)

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* Prior radiotherapy to less than 25% of bone marrow allowed provided the irradiated area is not the only site of measurable disease
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Other

* At least 3 weeks since prior therapy for cancer
* More than 4 weeks since prior investigational agents
* No other concurrent experimental medications
* No other concurrent therapy for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-10; Primary Completion 2005-08 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Survival | Patients are followed monthly for 3 months, every 2 months for 6 months, and then every 3 months thereafter

SECONDARY OUTCOMES:
Response rate (partial and complete response) | Patients are followed monthly for 3 months, every 2 months for 6 months, and then every 3 months thereafter
Time to progression | treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression.
Toxicity as measured by NCI CTC | at baseline and at the end of each course not at day 8
Quality of life as measured by the lung cancer symptom scale | At baseline, at restaging, before courses 2-6 of docetaxel*, and then at 1 and 3 months after study treatment. Arm II, QOL is assessed every 3 weeks until first disease progression and then before courses 2-6 of docetaxel.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Levitan, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States